CLINICAL TRIAL: NCT01677507
Title: Aqueous Humor Dynamic Components That Determine Intraocular Pressure Variance
Brief Title: Glaucoma Biomarkers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: University of Nebraska (Other); Mayo Clinic (Other); National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, Sayoko E. Moroi, PI, University of Michigan
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HUM00052276; R01EY022124 (NIH)
Record Dates: First submitted 2012-08-07; First posted 2012-09-03 (Estimated); Results first posted 2017-09-13 (Actual); Last update posted 2017-09-13 (Actual); Status verified 2017-08

CONDITIONS: Glaucoma; Healthy
Keywords: glaucoma; aqueous humor dynamics; intraocular pressure
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- timolol (Experimental): To compare the variation in response to timolol between individuals
  Interventions: Drug: Variation in eye pressure response to timolol and latanoprost treatment
- latanoprost (Active Comparator): To compare the variation in response to latanoprost between individuals
  Interventions: Drug: Variation in eye pressure response to timolol and latanoprost treatment

INTERVENTIONS:
Drug: Variation in eye pressure response to timolol and latanoprost treatment — Arm 1 is to test for variation in eye pressure response to timolol. Arm 2 is to test for variation in eye pressure response to latanoprost.

SUMMARY:
Glaucoma is a major cause of blindness. The inability to predict a patient's IOP response to medications is a critical barrier for the clinician to consistently provide highly effective IOP-based treatments. Current trial-and error approaches to glaucoma management are inefficient and have not addressed this barrier as there are no predictive factors for drug response. Our long-term goal is to improve outcomes by identifying biomarkers and environmental factors that profile a patient at risk for glaucoma by age-of-onset, rate of disease progression, "poor response" to treatment, and large IOP fluctuation. Our purpose of this research project is to address this critical barrier by focusing on physiological factors that predict IOP response to drugs.

ELIGIBILITY:
Inclusion Criteria:

* Either gender.
* Any self-declared ethnoracial category.
* Greater than or equal to 40 years.
* Healthy eyes with the crystalline lens, without glaucoma (cup:disc ratio < 0.8 both eyes; asymmetry of cup:disc ratio between eyes < 0.2).
* Open angles.
* Ability to cooperate for aqueous humor dynamic studies.
* Nonprescription and prescription topical ophthalmic products and systemic medications other than those mentioned in the exclusion criteria will be allowed during the study.
* Contact lenses removed prior to topical fluorescein instillation, and not used until the end of each fluorophotometry session.
* Able to participate on site over the multi-visit study period.

Exclusion Criteria:

* Women who are pregnant due to IOP changes.
* Any form of glaucoma, including extremely narrow angle with complete or partial closure.
* Current use of any glaucoma medication, either topically or orally.
* Chronic or recurrent inflammatory eye disease.
* Ocular trauma within the past 6 months.
* Ocular infection or ocular inflammation in the past 3 months.
* Clinically significant retinal disease.
* Any abnormality preventing reliable fluorophotometry of either eye, such as corneal scarring or severe dry eye that results in punctate fluorescein staining of the cornea.
* Intraocular surgery within 6 months.
* Serious hypersensitivity to any components of the study medications or risk from treatment with glaucoma medications, such as severe asthma or emphysema.
* Subjects must be on a stable regimen for at least 30 days prior to the Visit 1 regarding a chronic systemic medication that may affect IOP (i.e., sympathomimetic agents, beta-blockers, alpha-adrenergic agonists, alpha-adrenergic blockers, calcium channel blockers, angiotensin converting enzyme inhibitors, etc.). Any change of such medication during the study period will result in exclusion.
* Use of any glucocorticoid by any route. Subject must be washed out of the glucocorticoid for at least 2 weeks before study entry.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2012-08; Primary Completion 2016-08-30 (Actual); Study Completion 2016-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sayoko E Moroi, MD, PhD, Principal Investigator — University of Michigan
Locations (3):
- United States (3):
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - University of Nebraska Medical Center, Omaha, Nebraska

REFERENCES:
- [Derived] Liu M, Reed DM, Fan S, Kazemi A, Gulati V, Sit AJ, Moroi SE, Toris CB. Assessing Agreement of Intraocular Pressure from Four Mechanistically Different Tonometers in the Eye Dynamics and Engineering Network Clinical Trial. Ophthalmol Glaucoma. 2025 Aug 11:S2589-4196(25)00157-7. doi: 10.1016/j.ogla.2025.07.010. Online ahead of print. PMID 40803602
- [Derived] Kolli A, Toris CB, Reed DM, Gilbert J, Sit AJ, Gulati V, Kazemi A, Fan S, Musch DC, Moroi SE. The Effects of Topical Timolol and Latanoprost on Calculated Ocular Perfusion Pressure in Nonglaucomatous Volunteers. J Ocul Pharmacol Ther. 2021 Dec;37(10):565-574. doi: 10.1089/jop.2021.0068. Epub 2021 Oct 4. PMID 34610254
- [Derived] Man X, Costa R, Ayres BM, Moroi SE. Acetazolamide-Induced Bilateral Ciliochoroidal Effusion Syndrome in Plateau Iris Configuration. Am J Ophthalmol Case Rep. 2016 Oct;3:14-17. doi: 10.1016/j.ajoc.2016.05.003. Epub 2016 May 17. PMID 29226268

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 135 consented. Prior to baseline measures: 4 were excluded for ineligibility; 6 withdrew consent fully prior to baseline measurements.
  After baseline measures: an additional 2 were excluded based on physician decision, and 2 withdrew for participant decision.
  Thus, 121 participants are included for period 1.
Groups:
- Timolol Followed by Latanoprost: To compare the variation in response to timolol between individuals
  Variation in eye pressure response to timolol and latanoprost treatment: Arm 1 initial period is to test for variation in eye pressure response to timolol 0.5%, then washout.
  Period 2 is to test for variation in eye pressure response to latanoprost 0.005%.
- Latanoprost Followed by Timolol: To compare the variation in response to latanoprost between individuals
  Variation in eye pressure response to timolol and latanoprost treatment:
  Arm 1 initial period is to test for variation in eye pressure response to latanoprost 0.005%, then washout.
  Period 2 is to test for variation in eye pressure response to timolol 0.5%.
Period: Initial Assignment
Arm/Group | Timolol Followed by Latanoprost | Latanoprost Followed by Timolol
Started | 63 | 58
Completed | 63 | 56
Not Completed | 0 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Protocol Violation | 0 | 1
Period: Second Assigment
Arm/Group | Timolol Followed by Latanoprost | Latanoprost Followed by Timolol
Started | 63 | 56
Completed | 60 | 51
Not Completed | 3 | 5
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Adverse Event | 1 | 3

BASELINE CHARACTERISTICS:
Population: In addition to the 119 participants who were randomized to actual treatment, the baseline population includes the 9 who came for full baseline measurements before they were excluded or chose to withdraw.
Groups:
- Baseline of Entire Population: Both arms are included because the study design was a cross over intent to treat with glaucoma medications. All participants were treated with both medications.
Arm/Group | Baseline of Entire Population
Number analyzed (Participants) | 125
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.1 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94
  Male | 31
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 107
  Asian | 2
  Hispanic | 3
  Black or African American | 12
  American Indian | 1
Region of Enrollment [Number; unit: participants]
  United States | 125
Intraocular pressure [Mean (Standard Deviation); unit: mmHg]
  Right eye | 14.4 (3.5)
  Left eye | 13.9 (3.5)
Aqueous humor flow [Mean (Standard Deviation); unit: microliters/min] — Population: There was missing aqueous flow data on 2 participants.
  microliters/min
    Right eye: number analyzed (Participants) | 123
    Right eye | 3.1 (1.2)
    Left eye: number analyzed (Participants) | 123
    Left eye | 2.9 (0.9)
Episcleral venous pressure [Mean (Standard Deviation); unit: mmHg] — Population: One site used a different method to measure episcleral venous pressure (n=29)
  mmHg
    Right eye: number analyzed (Participants) | 96
    Right eye | 8.3 (1.7)
    Left eye | 7.9 (1.5)

OUTCOME MEASURES:

1. Primary Outcome: Variation in Eye Pressure Between Individuals.
Description: Eye pressure is a steady state quantitative trait that is measured in mm Hg. Eye pressure is determined by the following physiological factors (units of measure): eye fluid or aqueous humor production (microliters/minute), aqueous humor outflow (microliters/minute), outflow resistance (microliters/minute/mm Hg) and venous pressure (mm Hg) of the eye. All of these physiological factors will be determined under baseline condition and under glaucoma drug treatment.
Time Frame: Measurement after 1 week of drug treatment
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Timolol: To characterize the response to timolol in all participants.
- Latanoprost: To characterize the response to latanoprost in all participants.
Arm/Group | Timolol | Latanoprost
Number analyzed (Participants) | 114 | 116
mmHg
  RIght Eyes | 11.5 (3.2) | 11.3 (3.2)
  Left Eyes | 11.0 (3.0) | 11.0 (2.9)
Statistical Analysis 1: Comparison: Timolol; Right Eye treated vs. untreated; Test type: Other; p = 0.0001, t-test, 2 sided; Actually these are 2 sided paired t-tests; Mean Difference (Final Values) = 2.8, 95% CI 2-sided [2.4 to 3.3]
Statistical Analysis 2: Comparison: Timolol; Left Eye treated vs. untreated; Test type: Other; p = 0.0001, t-test, 2 sided; paired t-test, 2 sided; Mean Difference (Final Values) = 2.8, 95% CI 2-sided [2.5 to 3.2]
Statistical Analysis 3: Comparison: Latanoprost; Right Eye treated vs. untreated; Test type: Other; p = 0.0001, t-test, 2 sided; paired t-test, 2 sided; Mean Difference (Final Values) = 3.0, 95% CI 2-sided [2.5 to 3.4]
Statistical Analysis 4: Comparison: Latanoprost; Left Eye, treated vs. untreated; Test type: Other; p = 0.0001, t-test, 2 sided; paired t-test, 2 sided; Mean Difference (Final Values) = 2.9, 95% CI 2-sided [2.5 to 3.3]

2. Secondary Outcome: Variation in Aqueous Flow Between Individuals.
Description: Aqueous flow production (microliters/minute) will be determined under baseline condition and under glaucoma drug treatment.
Time Frame: 1 week after treatment
Population: These measurements can be difficult for participants to tolerate, so sometimes values are missing.
Measure: Mean (Standard Deviation); unit: microliters/min
Groups:
- Timolol: All participants while on timolol and during a post-timolol washout
- Latanoprost: All participants while on latanoprost and during a post-latanoprost washout
Arm/Group | Timolol | Latanoprost
Number analyzed (Participants) | 112 | 114
microliters/min
  Right eye: number analyzed (Participants) | 112 | 113
  Right eye | 1.9 (0.6) | 2.8 (0.9)
  Left eye: number analyzed (Participants) | 111 | 114
  Left eye | 2.0 (0.6) | 3.0 (1.0)
Statistical Analysis 1: Comparison: Timolol; Right Eye treated to untreated; Test type: Other; p = 0.0001, t-test, 2 sided; paired t test, 2 sided; Median Difference (Final Values) = 1.1, 95% CI 2-sided [0.9 to 1.3]
Statistical Analysis 2: Comparison: Timolol; Left Eye, treated vs. untreated; Test type: Other; p = 0.0001, t-test, 2 sided; paired t test, 2 sided; Median Difference (Final Values) = 0.9, 95% CI 2-sided [0.7 to 1.1]
Statistical Analysis 3: Comparison: Latanoprost; Right Eye, treated vs. untreated; Test type: Other; p = 0.94, t-test, 2 sided; paired t-test; Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-0.2 to 0.2]
Statistical Analysis 4: Comparison: Latanoprost; Left Eye, treated vs. untreated; Test type: Other; p = 0.54, t-test, 2 sided; paired t-test, 2 sided; Mean Difference (Final Values) = 0.05, 95% CI 2-sided [-0.1 to 0.2]

3. Secondary Outcome: Variation in Episcleral Venous Pressure.
Description: Episcleral venous pressure (mm Hg) of the eye will be determined under baseline condition and under glaucoma drug treatment.
Time Frame: 1 week treatment
Population: These measures can be difficult to obtain, so sometimes participants do not tolerate it and some values are missing.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Timolol | Latanoprost
Number analyzed (Participants) | 110 | 107
mmHg
  Right eye | 7.6 (1.5) | 7.7 (1.9)
  Left eye | 7.3 (1.5) | 7.4 (1.7)
Statistical Analysis 1: Comparison: Timolol; Right Eye, treated vs. untreated; Test type: Other; p = 0.04, t-test, 2 sided; paired t-test, 2 sided; Mean Difference (Final Values) = 0.4, 95% CI 2-sided [0.01 to 0.7]
Statistical Analysis 2: Comparison: Timolol; Left eye, treated vs. untreated; Test type: Other; p = 0.15, t-test, 2 sided; paired t-test, 2 sided; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-0.1 to 0.6]
Statistical Analysis 3: Comparison: Latanoprost; Right Eye, treated vs. untreated; Test type: Other; p = 0.52, t-test, 2 sided; paired t-test, 2 sided; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.3 to 0.6]
Statistical Analysis 4: Comparison: Latanoprost; Left Eye, treated vs. untreated; Test type: Other; p = 0.88, t-test, 2 sided; paired t-test, 2 sided; Mean Difference (Final Values) = 0.03, 95% CI 2-sided [-0.4 to 0.4]

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | Timolol | Latanoprost
All-Cause Mortality (participants affected / at risk) | 0/119 | 0/121
Serious Adverse Events (participants affected / at risk) | 0/119 | 0/121
Other Adverse Events (participants affected / at risk) | 0/119 | 0/121

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes